CLINICAL TRIAL: NCT05764304
Title: Therapeutic Evaluation of Treatment With Sinomenine Versus Glucocorticoid for Early Knee Osteoarthritis: A Prospective, Double-Blind, Randomized, Multicenter Clinical Trial
Brief Title: Sinomenine Versus Glucocorticoid for Knee OA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Changqing Zhang, Principal Investigator, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-277
Record Dates: First submitted 2023-02-17; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — sinomenine; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinomenine (Experimental)
  Interventions: Drug: Sinomenine
- Glucocorticoid (Active Comparator)
  Interventions: Drug: Glucocorticoid

INTERVENTIONS:
Drug: Sinomenine — Participants will receive one intra-articular injection every 4 months
  Arms: Sinomenine
Drug: Glucocorticoid — Participants will receive one intra-articular injection every 4 months
  Arms: Glucocorticoid

SUMMARY:
Both glucocorticoid and sinomenine are widely used in the routine clinical treatment of osteoarthritis, but there is still a lack of high level of clinical evidence for the direct comparison of efficacy between the two drugs. This trial aims to evaluate whether intraarticular injection of sinomenine was noninferior to intraarticular injection of glucocorticoid for symptom relief in patients with early knee arthritis, and whether intraarticular injection of sinomenine was superior to intraarticular injection of glucocorticoid for changes in tibial cartilage volume (measured by mean thickness) from baseline compared with intraarticular injection of glucocorticoid. 326 people will participate in the study at 3 different research/medical institutions, with centres competing for inclusion. This trial was designed by random blind method. This trial will last for 2 years and participants will receive 6 injections every 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 40 and <70.
2. Bilateral knee pain lasting for more than 6 months and most of the last month;
3. X-rays showed that Kellgren and Lawrence had grade 2 or 3 knee osteoarthritis.

Exclusion Criteria:

1. Kellgren and Lawrence Level 1 or 4.
2. Radiographs showed that the reduction of the lateral joint space was greater than or equal to the medial joint space.
3. The affected knee had been injected with glucocorticoid or hyaluronic acid within the past 6 months.
4. Have had knee surgery or plan to have joint surgery on the affected knee.
5. Other medical conditions such as: systemic or inflammatory joint diseases (rheumatoid arthritis), history of crystalline or neurological joints, other muscular, joint or nervous system diseases affecting lower limb function.
6. Have a needle phobia.
7. Immunosuppression or acute infection is present.
8. Patients are allergic to the drugs involved in the study.
9. Have or have had cancer or tumours.
10. Have a hemorrhagic disease or are receiving anticoagulant or antiplatelet therapy.
11. History of hyperlipidemia, or plasma total cholesterol ≥6.2mmol/L and triglycerides >2.3mmol/L
12. Have any other medical conditions that do not participate in the study, including contraindications to MRI, such as pacemakers.
13. Pregnancy.
14. Body mass Index (BMI) > 40 kg/m2.
15. Unable to attend all study appointments within 24 months;
16. Inability to understand written and spoken Chinese.
17. Any history of mental and psychological illness.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
total WOMAC score and tibial cartilage volume | 24 months after the first injection
  24 months after the first injection (1) the change in the total WOMAC score from baseline and whether sinomenine was noninferior to glucocorticoid, and (2) the change in tibial cartilage volume from baseline (on average thickness in mm) and whether sinomenine was noninferior to glucocorticoid.

SECONDARY OUTCOMES:
The Timed Up and Go and 20m walking time | 24 months after the first injection
  24 months after the first injection (1) the change in time from baseline in The Timed Up and Go (TUG) test and whether sinomenine was noninferior to glucocorticoid, and (2) the change in time spent at 20m walking time from baseline was and whether sinomenine was noninferior to glucocorticoid.

OTHER OUTCOMES:
Bone marrow lesion (BML) | 12 and 24 months after the first injection
  12 and 24 months after the first injection, to evaluate bone marrow lesion (BML) size of patients and whether sinomenine was noninferior to glucocorticoid.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang X, Lin Z, Lv M, Lu C, Hu B, Yu W, Wang Z, Liu X, Zhang C, Wu D, He Y. Cartilage organoids bridging bench to bedside: A steroid-free strategy for early osteoarthritis repair. Mater Today Bio. 2025 Dec 21;36:102688. doi: 10.1016/j.mtbio.2025.102688. eCollection 2026 Feb. PMID 41560786